CLINICAL TRIAL: NCT00600548
Title: Clinical Trial to Assess Efficacy and Safety of Orally Administered Miltefosine in Brazilian Patients With Cutaneous Leishmaniasis Compared to the Standard Care as Active Control
Brief Title: Trial of Miltefosine in Cutaneous Leishmaniasis (Brazil)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hospital Universitário Professor Edgard Santos (Other)
Collaborators: Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government); Ministerio de Ciencia e Innovación, Spain (Other Government); Ministry of Health, Brazil (Other Government); AEterna Zentaris (Industry)
Responsible Party: Paulo Roberto Lima Machado, Universidade Federal da Bahia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D-18506; 410559/2006-7
Record Dates: First submitted 2008-01-02; First posted 2008-01-25 (Estimated); Last update posted 2010-04-15 (Estimated); Status verified 2010-03

CONDITIONS: Treatment of Cutaneous Leishmaniasis in Brazil.
Keywords: Cutaneous leishmaniasis; Miltefosine; Meglumine antimoniate; L. braziliensis, L. guyanensis
MeSH Terms: conditions — Leishmaniasis, Cutaneous | interventions — miltefosine; Meglumine Antimoniate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1.1 (Experimental): Cutaneous leishmaniasis patients in Manaus-Amazonas randomized to receive Miltefosine.
  Interventions: Drug: Miltefosine.
- 1.2 (Active Comparator): Cutaneous leishmaniasis patients in Manaus-Amazonas randomized to receive Meglumine antimoniate (standard treatment).
  Interventions: Drug: Meglumine antimoniate.
- 2.1 (Experimental): Cutaneous leishmaniasis patients in Corte de Pedra-Bahia randomized to receive Miltefosine.
  Interventions: Drug: Miltefosine.
- 2.2 (Active Comparator): Cutaneous leishmaniasis patients in Corte de Pedra-Bahia randomized to receive Meglumine antimoniate (standard treatment).
  Interventions: Drug: Meglumine antimoniate.

INTERVENTIONS:
Drug: Miltefosine. — Miltefosine: Capsules containing 10 mg or 50 mg miltefosine; administered orally for 28 days at dosage of 2.5 mg/kg body weight per day.
  Other Names: Impavido.
  Arms: 1.1
Drug: Meglumine antimoniate. — Meglumine antimoniate administered by intravenous route for 20 days at the dosage of 20mg/kg/day.
  Other Names: Glucantime.
  Arms: 1.2
Drug: Miltefosine. — Miltefosine: Capsules containing 10 mg or 50 mg miltefosine; administered orally for 28 days at dosage of 2.5 mg/kg body weight per day.
  Other Names: Impavido.
  Arms: 2.1
Drug: Meglumine antimoniate. — Meglumine antimoniate administered by intravenous route for 20 days at the dosage of 20mg/kg/day.
  Other Names: Glucantime.
  Arms: 2.2

SUMMARY:
The hypothesis of this trial is that the therapeutic activity and safety of oral miltefosine in Brazilian patients with cutaneous leishmaniasis is similar or superior to the intravenous standard treatment (meglumine antimoniate - Glucantime®).

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed (untreated) cutaneous leishmaniasis with localized lesions and visualization of amastigotes in tissue samples or a positive culture or diagnosed by polymerase chain reaction (PCR) methods or by intradermal skin testing (Montenegro test).
* Number of lesions: 1 to 5 ulcerative lesions.
* Lesion´s diameter: 1 to 5 cm.
* Disease duration: up to three months.

Exclusion Criteria:

Safety concerns:

* Thrombocyte count <30 x 109/l
* Leukocyte count <1 x 109/l
* Hemoglobin <5 g/100 ml
* ASAT, ALAT, AP >3 times upper limit of normal range
* Bilirubin >2 times upper limit of normal range
* Serum creatinine or BUN >1.5 times upper limit of normal range
* Evidence of serious underlying disease (cardiac, renal, hepatic or pulmonary)
* Immunodeficiency or antibody to HIV
* Any non-compensated or uncontrolled condition, such as active tuberculosis, malignant disease, severe malaria, HIV, or other major infectious diseases
* Lactation, pregnancy (to be determined by adequate test) or inadequate contraception in females of childbearing potential for treatment period plus 2 months

Lack of suitability for the trial:

* Negative parasitology (aspirate/smear)or negative Montenegro test
* Any history of prior anti-leishmania therapy
* Any condition which compromises ability to comply with the study procedures
* Concomitant serious infection other than cutaneous

Administrative reasons:

* Lack of ability or willingness to give informed consent (patient and/or parent / legal representative)
* Anticipated non-availability for study visits/procedures

Ages: 2 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2007-07; Primary Completion 2009-03 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Cure rate or complete cicatrization of the ulcer. | 6 months after treatment.
  Bidirectional measurements of ulcers will be taken of the patients' lesions at the initial visit, and at each follow-up visit with standardized caliper. The area involved will be calculated as the product of the two measurements.
  All lesions will be categorized as either active or healed (cured) at follow-up visits. Only lesions with complete re-epithelialization, without raised borders, infiltrations or crusts will be considered healed. Evaluation of the lesions will be performed by 2 clinicians who will be unaware of the group assignment of all patients.

SECONDARY OUTCOMES:
Inicial cure rate or complete cicatrization of the ulcer. | 2 months after treatment.
  Bidirectional measurements of ulcers will be taken of the patients' lesions at the initial visit, and at each follow-up visit with standardized caliper. The area involved will be calculated as the product of the two measurements.
  All lesions will be categorized as either active or healed (cured) at follow-up visits. Only lesions with complete re-epithelialization, without raised borders, infiltrations or crusts will be considered healed. Evaluation of the lesions will be performed by 2 clinicians who will be unaware of the group assignment of all patients.

CONTACTS AND LOCATIONS:
Overall Officials: Paulo RL Machado, MD, PhD, Principal Investigator — Federal University of Bahia
Locations (2):
- Brazil (2):
  - Fundação de Medicina Tropical do Amazonas, Manaus, Amazonas
  - Posto de Saúde de Corte de Pedra, Tancredo Neto, Estado de Bahia

REFERENCES:
- [Derived] Machado PR, Ampuero J, Guimaraes LH, Villasboas L, Rocha AT, Schriefer A, Sousa RS, Talhari A, Penna G, Carvalho EM. Miltefosine in the treatment of cutaneous leishmaniasis caused by Leishmania braziliensis in Brazil: a randomized and controlled trial. PLoS Negl Trop Dis. 2010 Dec 21;4(12):e912. doi: 10.1371/journal.pntd.0000912. PMID 21200420